CLINICAL TRIAL: NCT07049965
Title: Clinical Profile of Appendicitis and Comparative Study for Use of Harmonic Scalpel (Seal and Cut) and Suture Ligation of Base of Appendix During Laparoscopic Appendectomy
Brief Title: Comparative Study of Harmonic Scalpel vs. Suture Ligation for Appendix Base During Laparoscopic Appendectomy
Acronym: HASSEL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GSVM Medical College (Other)
Responsible Party: Principal Investigator, Apoorva Mathur, Principal investigator, Junior Resident, Department of General Surgery, GSVM Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/BMHR/2024/35
Record Dates: First submitted 2025-06-18; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Appendicitis
Keywords: Laparoscopic appendicectomy; Harmonic scalpel; Suture ligation; Surgical site infection; Operative time; Appendicitis; Appendiceal stump closure
MeSH Terms: conditions — Appendicitis; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Group, Active controlled trial Computer generated randomisation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Suture ligation (Active Comparator): Participants will undergo laparoscopic appendectomy where the base of the appendix is secured using conventional intracorporeal suture ligation, using absorbable sutures.
  Interventions: Procedure: Suture ligation
- Harmonic Scalpel (Experimental): Participants in this group will undergo laparoscopic appendectomy in which the base of the appendix is sealed and divided using a harmonic scalpel. The device simultaneously cuts and coagulates tissue using ultrasonic energy, potentially reducing operative time, blood loss, and thermal injury compared to conventional methods.
  Interventions: Device: Harmonic Scalpel

INTERVENTIONS:
Procedure: Suture ligation — Participants will undergo laparoscopic appendectomy in which the base of the appendix is ligated using intracorporeal suturing with absorbable material. This is the conventional technique used to prevent stump leakage.
  Arms: Suture ligation
Device: Harmonic Scalpel — Participants will undergo laparoscopic appendectomy where the base of the appendix is sealed and divided using the harmonic scalpel. This ultrasonic energy-based device cuts and coagulates tissue simultaneously, potentially reducing operative time and blood loss.
  Arms: Harmonic Scalpel

SUMMARY:
This study is a comparative study between use of suture ligation vs harmonic scalpel for sealing and cutting the base of appendix.

The ideal method for closing the appendix stump should be safe, reliable, simple to use, and cost-effective. Various techniques have been introduced for this purpose, each with its advantages and disadvantages. However, no clear consensus has been reached in the literature regarding which technique is superior.

This study is to compare the two groups in terms of operative time and postoperative complications and to reach a conclusion as to which one of the two is superior.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common causes of emergency abdominal surgery worldwide. Laparoscopic appendectomy has become the standard of care due to its advantages of faster recovery and reduced postoperative complications. A key step in the procedure is the secure closure of the base of the appendix to prevent intra-abdominal leakage and stump complications. Traditionally, this is done using intracorporeal suture ligation or endoloops. However, the introduction of energy devices such as the harmonic scalpel has offered a potential alternative that combines cutting and coagulation, potentially reducing operative time and simplifying the procedure.

This prospective interventional study aims to compare the effectiveness and safety of harmonic scalpel (seal-and-cut technique) versus conventional suture ligation for closure of the appendix base during laparoscopic appendectomy in patients with uncomplicated acute appendicitis. A total of 60 patients will be enrolled and randomized into two groups: Group A (Harmonic Scalpel) and Group B (Suture Ligation). Both groups will undergo standard laparoscopic appendectomy with the only variable being the method of securing the appendix stump.

The primary outcomes of interest include operative time,Postoperative leak, Postoperative ileus,Surgical site infection and Hospital Stay and secondary outcome of interest include Recovery and Postoperative complications. Follow-up will be done on postoperative day 1, day 7, day 30 and 3 months. This study seeks to determine whether the harmonic scalpel offers a safe and effective alternative to conventional ligation, potentially simplifying surgical technique and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 5 - 65 years
2. Any gender
3. Patient willing to undergo laparoscopic appendectomy
4. Acute appendicitis confirmed by clinical and radiological analysis
5. Alvarado Score ≥7
6. Alvarado Score ≥5 with positive ultrasound findings

Exclusion Criteria:

1. Patient with base of appendix highly inflamed / gangrenous
2. Any other intra-abdominal pathology other than acute appendicitis, e.g., appendicular mass, appendicular abscess, tuberculosis, carcinoid tumor, pelvic inflammatory disease, ovarian tumors, ceacal mass, etc.
3. Patients declared unfit for laparoscopic surgery during preoperative assessment
4. Patients having severe co morbid condition - COPD/CAD/CHF

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative( measured during surgical procedure on day 1)
  Total duration of surgery in minutes, measured from skin incision to completion of appendix base closure. Used to compare efficiency between harmonic scalpel and suture ligation techniques.

SECONDARY OUTCOMES:
Position of appendix | Intraoperative ( day 1)
  Anatomical position of the appendix (e.g., retrocecal, pelvic, subhepatic) recorded intraoperatively to assess distribution and influence on technical difficulty or operative time.
Postoperative Leak | Upto 7 days post-operation
  Presence of intra-abdominal fluid collection or fecal contamination diagnosed clinically or via imaging, indicating leak from the appendix stump.
Postoperative Ileus | Upto 5 days post-operation
  Delayed return of bowel function defined by absence of flatus or bowel movements, abdominal distension, or need for nasogastric decompression.
Surgical site infection | Up to 30 days post-operation
  Superficial or deep wound infection including erythema, discharge, or wound dehiscence.
Hospital stay | From date of surgery until discharge, assessed upto 14 days
  Total number of days from the date of operation to discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Apoorva Mathur, MBBS, Principal Investigator — Ganesh Shankar Vidhyarthi Memorial Medical College Kanpur
Locations (1):
- Ganesh Shankar Vidhyarthi Memorial Medical College Kanpur, Kanpur, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to operative time, hospital stay, and postoperative complications
Supporting Information: CSR
Time Frame: 6 months after publication of results for 2 years
Access Criteria: Qualified researchers upon reasonable request

DOCUMENTS (1):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT07049965/Prot_000.pdf